CLINICAL TRIAL: NCT03321773
Title: Compare 14-day Reverse Hybrid Therapy and 14-day Triple Therapy Plus Bismuth on Helicobacter Pylori Eradication
Brief Title: Comparing the Efficacy of 14-day Reverse Hybrid Therapy and 14-day Triple Therapy Plus Bismuth Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Feng-Woei Tsay, Assistant Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS16-CT10-17
Record Dates: First submitted 2017-10-20; First posted 2017-10-26 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication rate
MeSH Terms: interventions — Pantoprazole; Amoxicillin; Clarithromycin; bismuth tripotassium dicitrate; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- triple therapy plus bismuth therapy (Experimental): pantoprazole 40mg twice daily for 14 days, amoxicillin 1g twice daily for 14 days, clarithromycin 500mg twice daily for 14 days, bismuth subcitrate 240mg twice daily for 14 days.
  Interventions: Drug: triple therapy plus bismuth therapy
- reverse hybrid therapy (Active Comparator): (pantoprazole 40mg twice daily for 7 days, amoxicillin 1 g twice dailyfor 7 days, clarithromycin 500 mg twice daily for 7 days, and metronidazole 500 mg twice daily for 7 days) followed by (pantoprazole 40mg twice daily for 7 days and amoxicillin 1 g twice daily for 7 days)
  Interventions: Drug: reverse hybrid therapy

INTERVENTIONS:
Drug: triple therapy plus bismuth therapy — pantoprazole 40mg twice daily for 14 days, amoxicillin 1g twice daily for 14 days, clarithromycin 500mg twice daily for 14 days, bismuth subcitrate 240mg twice daily for 14 days.
  Other Names: pantoprazole 40 mg; amoxicillin 1g; clarithromycin 500mg; bismuth subcitrate 240mg
  Arms: triple therapy plus bismuth therapy
Drug: reverse hybrid therapy — (pantoprazole 40mg twice daily for 7 days, amoxicillin 1 g twice dailyfor 7 days, clarithromycin 500 mg twice daily for 7 days, and metronidazole 500 mg twice daily for 7 days) followed by (pantoprazole 40mg twice daily for 7 days and amoxicillin 1 g twice daily for 7 days)
  Other Names: pantoprazole 40mg; amoxicillin 1g; clarithromycin 500mg; metronidazole 500mg
  Arms: reverse hybrid therapy

SUMMARY:
Reverse hybrid therapy achieves a higher eradication rate than bismuth (triple therapy plus bismuth) remains unanswered

DETAILED DESCRIPTION:
With the rising prevalence of antimicrobial resistance, the failure rate of the 7-day standard triple therapy has declined to unacceptable level (<80%) worldwide. Several regimens were suggested to replace standard triple therapy in the area with high clarithromycin resistance, including sequential therapy, concomitant therapy, hybrid therapy and bismuth containing quadruple therapy. A 14-day hybrid therapy invented by our study group appears very promising in H. pylori eradication, achieving eradication rates of 95%. A clinical trial by Hsu et al from our hospital showed 12-day reverse hybrid therapy also achieved high eradication rate, and improved the compliance of patients. Even prolong the treatment duration of standard triple therapy from 7 days to 12 days, the efficacy of eradication was still < 90% (85-88%). The limitation of triple therapy in against resistant-stains was still existed. The addition of bismuth (triple therapy plus bismuth) can improve cure rates despite a high prevalence of antimicrobial resistance. The major bismuth effect is to add an additional 30%-40% to the success with resistant infections. However the direct compare the efficacy between 14-day reverse hybrid therapy and 14-day triple therapy plus bismuth is still insufficiency in Taiwan and worldwide. Choosing a navel therapy or a modifying triple therapy can get better efficacy, it is remained to be determined. Besides genotyping polymorphism of CYP2C19 influenced the metabolism of proton pump inhibit, and could cause decreasing of eradication rate of standard triple therapy. But the influence in 14-day reverse hybrid therapy and 14-day triple therapy plus bismuth is unclear.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H pylori-infected outpatients, at least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H pylori-eradication therapy
* ingestion of antibiotics or bismuth within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants in Which H. Pylori Was Eradicated | sixth week after the end of anti- H. pylori therapy
  To assess eradication efficacy,repeated endoscopy with rapid urease test, histological examination and culture or Urea breath test.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Woei Tsay, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan